CLINICAL TRIAL: NCT07306117
Title: A Person-centered, Theory-based, Intervention to Enhance Adolescents' Motivation for Adequate Oral Hygiene Behavior - Method Development Through the Integration of Digital Technology.
Brief Title: A Person-centered, Theory-based, Intervention - Method Development Through the Integration of Digital Technology.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Sandra Lod Dimenäs, Principal investigator, Göteborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dnr: 2025-06217-01
Record Dates: First submitted 2025-12-04; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis
Keywords: Qualitative study; Gingivitis; Plaque; prevention; periodontal disease; behavioral change intervention; person-centered care; behavioral medicine; adolescents; oral health; oral hygiene; qualitative interviews
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Periodontal Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Adolescents will be treated in accordance with the person-centered and theory-based intervention (based on social cognitive theory and including the behavioral change techniques goal setting, planing and self-monitoring) that was tested/evaluated in the previous treatment study, but where the written diary for self-monitoring of oral hygiene behavior is replaced by a mobile health application. The application is intended to be used for self-monitoring during the active/initial phase of the behavioral intervention, which includes two physical and one digital visit over 12 weeks, followed by a follow-up/evaluation visit at six months. In addition, after completion of the initial intervention phase, the adolescents will be offered a person-centered digital maintenance meeting as support to promote/maintain positive oral health/oral hygiene habits. The maintenance phase covers the period from six to twelve months when the treatment in the pilot study ends.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person-centered, theory-based, intervention (Experimental): This treatment is the most recommended when behavioral change is needed to promote adequate oral hygiene - based on the Swedish National Guidelines for Dental Care (National Board of Health and Welfare, 2022). The aim is to, with a qualitative approach, explore views on the health application for self-monitoring and supportive person-centered digital maintenance meetings to promote new/positive oral hygiene habits.
  Interventions: Behavioral: Person-centered, theory-based, intervention

INTERVENTIONS:
Behavioral: Person-centered, theory-based, intervention — The person-centered intervention is based on theory of health behavior and includes behavior change techniques (personal goal setting for oral hygiene and oral health, planning, and monitoring of behavior). The dental hygienists use a collaborative communication method inspired by motivational interviewing. This intervention is the most recommended treatment for behavior change in cases of unhealthy lifestyle habits according to the National Guidelines for Dental Care (The National Board of Health and Welfare, 2022).
  The initial intervention phase includes three visits:
  Visit 1 (Baseline) - face-to-face (approx. 60 min) Visit 2 (2-3 weeks after baseline) - face-to-face (approx. 40 min) Visit 3 (10-12 weeks after baseline) - digital (approx. 30 min)
  After 6 months, a follow-up is conducted (Visit 4 - face-to-face, approx. 40 min). Between 6 and 12 months (maintenance phase), one digital meeting is offered to support maintenance of new/positive oral hygiene habits.

SUMMARY:
Studies have shown that Swedish adolescents have poor oral hygiene and with high prevalence of gingivitis. Therefore, more effective preventive programs in dental care are needed. The project aims to examine whether a health application and follow-up person-centered digital meetings can serve as support in person-centered and theory-based behavioral interventions to promote and maintain positive oral health habits.

DETAILED DESCRIPTION:
Specific Aim - Purpose:

The overarching aim of the project is to develop more effective preventive programs targeting adolescents to promote oral/periodontal health.

Within the framework of the project, a clinical treatment study was recently conducted in which the investigators tested a person-centered, theory-based, behavioral intervention to strengthen adolescents' motivation for adequate oral hygiene behavior. The present study is a continuation of the project, focusing on method development of the intervention through the introduction of digital technology:

The specific aim of the present study is to:

* test a mobile health application as support/tool in person-centered, theory-based, interventions targeting young people in dental care, and
* explore whether person-centered digital maintenance meetings can be perceived as supportive for maintaining/promoting positive oral health/oral hygiene habits over time.

Background:

In Sweden, all children and adolescents are included in preventive programs within the free-of-charge dental care. Despite this, epidemiological studies show that adolescents have remarkably poor oral hygiene with a high prevalence of gingivitis. Gingivitis is a reversible condition, but if left untreated it can develop into chronic and destructive periodontitis. The prevalence of periodontitis is about 40% in the adult population, with associated consequences and significant costs for treatment/rehabilitation. The most important factor in preventing disease progression is establishing infection control through adequate daily oral hygiene. Dental professionals play a key role in educating and strengthening the individual's motivation for such health-promoting behavior.

Previous epidemiological studies have identified individual and environmental factors that interact with adolescents' health behavior and periodontal health status. When meeting young patients, it is important for dental professionals to consider such factors for a person-centered approach in interventions aimed at promoting health behaviors. Studies within dentistry indicate that behavioral interventions are more effective when based on theories of health behavior compared to conventional information/instruction in the treatment of adults with periodontitis. A systematic review concluded that key components of such theory-based interventions were that the individual:

(i) formulates personal goals for oral health and health behavior, (ii) plans for the implementation of the behavior in question, and (iii) monitors their behavior through self-monitoring (diary).

Furthermore, for positive behavior change to occur, it is crucial that the individual has knowledge and insight into their disease and understands the personal benefits of adopting a more health-oriented behavior. The use of a person-centered and collaborative communication method, such as motivational interviewing, by dental professionals also appears to be important in interventions aimed at improving oral health/oral hygiene behavior. However, there is a need for more studies in this area, including studies that do not only involve adult patients with periodontitis but also other patient/age groups. The importance of studies conducted in general dental practice has also been emphasized.

Based on knowledge generated in our own and others' studies, as described above, a randomized clinical field study was planned and conducted to test the effect of a person-centered, theory-based, intervention targeting adolescents to increase motivation for periodontal infection control, i.e., adequate oral hygiene behavior. The study included 312 adolescents (16-17 years), who were treated by dental hygienists (DH) in general dental care, Public Dental Service, Region Västra Götaland. The person-centered, theory-based intervention included components such as goal setting, planning, and self-monitoring of oral hygiene behavior, and DHs used motivational interviewing skills in communication (for further details see: ClinTrials.gov NCT02906098). Evaluation/results at six months showed that the person-centered, theory-based intervention (test) was more effective in establishing periodontal infection control compared to conventional information/instruction (control). In follow-up qualitative interviews with adolescents, feedback was provided on components of the test intervention that were perceived as working well and what could be improved. One finding from these interviews was that the written diary used by adolescents for self-monitoring of oral hygiene behavior was perceived as "old-fashioned" and difficult to keep track of, which meant that the diary was not always used as intended. Adolescents stated during interviews that they understood the benefit of the diary but that a mobile/smartphone application for self-monitoring could be an alternative that better suited their lives and needs. The use of smartphone applications has become an integral part of young people's lives, and there is growing interest in using such applications in interventions focused on behavioral change, but few studies have so far used such technology in interventions aimed at improving oral health habits. Furthermore, interviews with adolescents who participated in the previous treatment study also revealed a need for continued support after the initial intervention phase, which ended after six months, to maintain newly acquired and more positive oral health/oral hygiene habits over time. Interviews with DHs who treated adolescents within the framework of the previous treatment study confirmed adolescents' need for continued support but were hesitant to offer more physical visits and suggested that follow-up digital meetings could be an alternative, which the investigator also intend to introduce and test within the framework of the present pilot study. The introduction of digital meetings as a complement to in-person visits is becoming increasingly common in healthcare, but no studies has tested this in relation to person-centered interventions focusing on adolescents' oral health.

Significance:

Within the free-of-charge dental care system for children and adolescents, substantial resources are invested in the prevention of oral diseases. It is, of course, of utmost importance to continuously evaluate the measures implemented in dental care and to develop and improve methods that promote good oral health over time. Epidemiological data highlight the need to develop more effective methods to increase adolescents' motivation for improved oral hygiene and thereby prevent periodontal disease progression. Considering the prevalence of periodontitis in the population and the consequences/costs associated with the disease, effective preventive measures are of great significance. Studies indicate that behavioral interventions are more effective when based on theory of health behavior. These studies have mainly included adult patients with periodontitis treated in specialist clinics. There is a need for studies that include young individuals/patients and studies conducted in general dental care. The present project therefore contribute essential knowledge for the design of more effective preventive programs targeting young individuals in general dental care. The project may also provide insights of value beyond the dental care field regarding how to influence adolescents toward health-promoting behaviors.

Materials & Methods:

The present study primarily adopts a qualitative methodological approach. The research team possesses solid expertise in qualitative methodology as well as other relevant knowledge and competencies necessary for the study's implementation.

Study Design and Participants:

Adolescents who, during a routine examination at the Public Dental Service, exhibit poor oral hygiene status (gingivitis and/or plaque on ≥50% of tooth surfaces) and who therefore are in need of individualized behavioral treatment will be informed about the study's purpose and asked if they are interested in participating. Approximately 25 patients/adolescents are planned to be included in the pilot study. These will be treated by five DHs (approximately five patients each) in accordance with the person-centered and theory-based intervention, but where the written diary for self-monitoring of oral hygiene behavior is replaced by a mobile health application. The application is intended to be used for self-monitoring during the active/initial phase of the behavioral intervention, which includes two physical and one digital visit over 12 weeks, followed by a follow-up/evaluation visit at six months. In addition, after completion of the initial intervention phase, the adolescents will be offered a person-centered digital maintenance meeting with their DH to promote/maintain positive oral health/oral hygiene habits. The maintenance phase covers the period from six to twelve months when the treatment in the pilot study ends.

Participating dental hygienists will undergo training prior to the study's implementation. During the implementation phase, a study coordinator will maintain regular contact with participating dental hygienists and provide support for any questions that may arise.

Data Collection & Analysis:

Data collection will be carried out through focus group interviews, but questionnaire-based and clinical data will also be collected at baseline.

Semi-structured focus group interviews (4-6 participants per group) will be conducted with current study participants (adolescents and treating DH, respectively) after 12 months, focusing on:

(i) the design/content and usability/usefulness of the application, and (ii) experiences/usefulness of digital maintenance meetings.

Questionnaire-based data will be collected from adolescents at study start/baseline. The questions focus on personal background characteristics, self-rated oral and general health, and oral hygiene behavior. The questionnaire will be completed by the adolescents in the waiting room before treatment and placed by themselves in a sealed envelope. The questions have been tested in previous studies among adolescents. Clinical data (plaque and bleeding) will be recorded by the treating DH at baseline. Questionnaire-based and clinical data will only be presented descriptively.

Data obtained through focus group interviews will be analyzed using qualitative content analysis. NVivo software will be used for data management. The analysis will be conducted in close collaboration among team members representing different professional and research fields (Oral Health, Psychology, Education, and Nursing Science with a particular focus on person-centered care).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (16-17 years)
* Gingivitis and/or plaque on ≥50% of tooth surfaces at dental examination.

Exclusion Criteria:

* Adolescents judged as not capable to understand the study information in order to make a considered choice about participation (The Swedish Ethical Review Act; SFS 2003:460, § 18).
* Adolescents with obvious difficulties with the Swedish language.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | 12 months after baseline.
  This pilot study has mainly a qualitative approach where the adolescents and the dental hygienists who provide the treatment will be interviewed regarding experiences and views on the health application for self-monitoring and supportive person-centered digital meetings.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L. Dimenäs, Odont. Dr, Principal Investigator — Departement of Periodontology, Institute of Odontology, University of Gothenburg
Locations (1):
- Folktandvården Västra Götaland, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] National Board of Health and Welfare (2022). Nationella riktlinjer för tandvård - stöd för styrning och ledning 2022 (in Swedish). Retrieved from https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/nationella-riktlinjer/2022-9-8114.pdf in September 2025. Information in English about the guidelines: https://www.socialstyrelsen.se/en/clinical-practise-guidelines-and-regulations/regulations-and-guidelines/national-guidelines/
- [Background] Ostberg AL, Ericsson JS, Wennstrom JL, Abrahamsson KH. Socio-economic and lifestyle factors in relation to priority of dental care in a Swedish adolescent population. Swed Dent J. 2010;34(2):87-94. PMID 20701217
- [Background] Werner H, Hakeberg M, Dahlstrom L, Eriksson M, Sjogren P, Strandell A, Svanberg T, Svensson L, Wide Boman U. Psychological Interventions for Poor Oral Health: A Systematic Review. J Dent Res. 2016 May;95(5):506-14. doi: 10.1177/0022034516628506. Epub 2016 Jan 29. PMID 26826109
- [Background] Wahlin A, Papias A, Jansson H, Norderyd O. Secular trends over 40 years of periodontal health and disease in individuals aged 20-80 years in Jonkoping, Sweden: Repeated cross-sectional studies. J Clin Periodontol. 2018 Sep;45(9):1016-1024. doi: 10.1111/jcpe.12978. Epub 2018 Jul 27. PMID 29971805
- [Background] Newton JT, Asimakopoulou K. Managing oral hygiene as a risk factor for periodontal disease: a systematic review of psychological approaches to behaviour change for improved plaque control in periodontal management. J Clin Periodontol. 2015 Apr;42 Suppl 16:S36-46. doi: 10.1111/jcpe.12356. PMID 25639708
- [Background] Ericsson JS, Wennstrom JL, Lindgren B, Petzold M, Ostberg AL, Abrahamsson KH. Health investment behaviours and oral/gingival health condition, a cross-sectional study among Swedish 19-year olds. Acta Odontol Scand. 2016;74(4):265-71. doi: 10.3109/00016357.2015.1112424. Epub 2015 Nov 24. PMID 26599291
- [Background] Ericsson JS, Ostberg AL, Wennstrom JL, Abrahamsson KH. Oral health-related perceptions, attitudes, and behavior in relation to oral hygiene conditions in an adolescent population. Eur J Oral Sci. 2012 Aug;120(4):335-41. doi: 10.1111/j.1600-0722.2012.00970.x. Epub 2012 Jun 25. PMID 22813224
- [Background] Ericsson JS, Abrahamsson KH, Ostberg AL, Hellstrom MK, Jonsson K, Wennstrom JL. Periodontal health status in Swedish adolescents: an epidemiological, cross-sectional study. Swed Dent J. 2009;33(3):131-9. PMID 19994563
- [Background] Dimenäs SL. Behavioral Intervention for Improved Oral Hygiene in Adolescents - A Person-Centered and Theory-Based Approach. 2024. PhD-thesis, University of Gothenburg, Sweden.
- [Background] Dimenas SL, Andersson JS, Jonsson B, Lundgren J, Petzold M, Ostberg AL, Abrahamsson KH. Adolescents' self-reported experiences following a person-centred, theory-based educational intervention versus conventional education for improved oral hygiene: Analysis of secondary outcomes of a randomized field study. J Clin Periodontol. 2024 Jan;51(1):63-73. doi: 10.1111/jcpe.13883. Epub 2023 Oct 11. PMID 37822115
- [Background] Dimenas SL, Jonsson B, Lundin M, Lundgren J, Abrahamsson KH. Changing from disease-centred to person-centred - Swedish dental hygienists' views on a theory-based behavioural intervention for improved oral hygiene among adolescents. Int J Dent Hyg. 2024 Nov;22(4):971-981. doi: 10.1111/idh.12811. Epub 2024 Apr 24. PMID 38659277
- [Background] Dimenas SL, Ostberg AL, Lundin M, Lundgren J, Abrahamsson KH. Adolescents' experiences of a theory-based behavioural intervention for improved oral hygiene: A qualitative interview study. Int J Dent Hyg. 2022 Nov;20(4):609-619. doi: 10.1111/idh.12606. Epub 2022 Aug 15. PMID 35925040
- [Background] Dimenas SL, Jonsson B, Andersson JS, Lundgren J, Petzold M, Abrahamsson I, Abrahamsson KH. A person-centred, theory-based, behavioural intervention programme for improved oral hygiene in adolescents: A randomized clinical field study. J Clin Periodontol. 2022 Apr;49(4):378-387. doi: 10.1111/jcpe.13601. Epub 2022 Feb 23. PMID 35132653
- [Background] Dimenäs SL. Smartphone-applikationer vid beteendeförändring: En litteraturstudie med fokus på interventioner i syfte att påverka unga individers hälsobeteende. Examensarbete för magister i Oral Hälsa, 15 hp. Göteborgs universitet, 2017
- [Background] Carra MC, Detzen L, Kitzmann J, Woelber JP, Ramseier CA, Bouchard P. Promoting behavioural changes to improve oral hygiene in patients with periodontal diseases: A systematic review. J Clin Periodontol. 2020 Jul;47 Suppl 22:72-89. doi: 10.1111/jcpe.13234. PMID 31912530
- [Background] Abrahamsson KH, Koch G, Norderyd O, Romao C, Wennstrom JL. Periodontal conditions in a Swedish city population of adolescents: a cross-sectional study. Swed Dent J. 2006;30(1):25-34. PMID 16708853